CLINICAL TRIAL: NCT01955226
Title: Unit Based Comparison of Non- Versus Chlorhexidine-Impregnated Central Line Dressings
Brief Title: CHG Dressings in Children With Central Lines
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Giuliano913
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Children With Central Venous Access

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tegaderm CHG clear dressing (Experimental): Patients randomized to receive Tegaderm CHG clear dressing. All central line care will remain uniform between the two groups as dictated by the central line maintenance bundle currently directing central line care in our children's hospital.
  Interventions: Other: Tegaderm CHG clear dressing
- Standard clear Tegaderm dressing (Active Comparator): Patients randomized to receive standard clear Tegaderm dressing. All central line care will remain uniform between the two groups as dictated by the central line maintenance bundle currently directing central line care in our children's hospital.
  Interventions: Other: Standard clear Tegaderm dressing

INTERVENTIONS:
Other: Tegaderm CHG clear dressing — Tegaderm CHG clear dressing will be used in central line care and will remain uniform as dictated by the central line maintenance bundle currently directing central line care in our children's hospital.
  Arms: Tegaderm CHG clear dressing
Other: Standard clear Tegaderm dressing — Standard clear Tegaderm dressing will be used in central line care and will remain uniform as dictated by the central line maintenance bundle currently directing central line care in our children's hospital.
  Arms: Standard clear Tegaderm dressing

SUMMARY:
The purpose of this study is to determine whether Tegaderm CHG clear dressing reduces the number of unscheduled central catheter dressing changes compared to standard clear Tegaderm IV dressing in pediatric patients between the ages of 2 months to 18 years with central venous access. Secondarily, we will monitor contact skin irritation and central line associated blood stream infections.

DETAILED DESCRIPTION:
In this prospective, randomized, cohort study, we plan on enrolling all patients 2 months to 18 years of age admitted with a central venous catheter expected to be in place for > 48 hours. Patients will be randomized to either receive 1) Tegaderm CHG clear dressing or 2) standard clear Tegaderm IV dressing. All central line care will remain uniform between the two groups as dictated by the central line maintenance bundle currently directing central line care in our children's hospital. Study completion will occur at the time of central line removal or discharge from the hospital, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* All patients 2 months to 18 years of age admitted with a central venous catheter expected to be in place for > 48 hours.

Exclusion Criteria:

* Patients with known allergies to chlorhexidine or Tegaderm and those previously enrolled in this study will be excluded.
* Patients with portacatheters

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction in unscheduled central catheter dressing changes | Study completion (Study completion will occur at the time of central line removal or discharge from the hospital, whichever comes first). On average 2 weeks.
  The policy at our institution is to change central catheter dressings every 7 days unless they are soiled or detached. We will document dressing changes for the duration of line use and document the reason for the dressing change.

SECONDARY OUTCOMES:
Blood Stream Infection | Discharge (at 2 weeks or more)
  Blood stream infections will be tallied and reported per 1,000 central line days. Infection is attributed to the line if a culture becomes positive when the line is in up to 48 hours after removal.
Skin irritation | Study completion (Study completion will occur at the time of central line removal or discharge from the hospital, whichever comes first). On average 2 weeks.
  Skin irritation will be assessed using the Scoring of patch tests according to the International Contact Dermatitis Research Group. Scores of 0 are defined as no irritation, 1/2-1+ as minor irritation whereas scores greater than or equal to 2+ will be classified as severe and will require dressing removal.
  The clinical team will photograph each central line insertion site with every dressing change and save the most severe skin irritation photo for analysis. These pictures will be sequentially numbered and a master list will link them to each patient.

CONTACTS AND LOCATIONS:
Overall Officials: John S Giuliano Jr, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States